CLINICAL TRIAL: NCT01254331
Title: Open Label, Multicenter, Trial to Evaluate Safety, Tolerability and Efficacy of Tocilizumab in Monotherapy or in Combination With MTX in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Current Non Biologic DMARDs
Brief Title: An Open-label Study With Tocilizumab in Patients With Rheumatoid Arthritis in a Local Environment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22642
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra] — tocilizumab 8 mg/kg intravenous infusion every 4 weeks for a total of 6 infusions

SUMMARY:
This open-label, multi-center study in a local environment will evaluate the safety and the effect on disease activity with regard to reduction in signs and symptoms over 6 months of treatment in patients with moderate to severe active rheumatoid arthritis who experienced an inadequate response to a non-biologic DMARD. Tocilizumab 8 mg/kg will be administered as an intravenous infusion every 4 weeks for a total of 6 infusions as monotherapy or in combination with methotrexate (MTX). The anticipated time of study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years of age
* Moderate to severe rheumatoid arthritis defined as DAS 28>3.2
* Body weight </=150 kg
* Patient on at least 1 non-biologic DMARD on a stable dose for at least 8 weeks at any time prior to study start
* Inadequate clinical response to a stable dose of a non-biologic DMARD

Exclusion Criteria:

* Major surgery within 8 weeks prior to screening or planned major surgery within 6 months following enrollment
* Rheumatic autoimmune disease other than rheumatoid arthritis (RA)
* Functional class IV as defined by the ACR classification
* History or current inflammatory joint disease other than RA
* Previous treatment with any cell depleting therapy
* Previous treatment with methotrexate
* Previous treatment with tocilizumab
* Previous treatment with any biologic drug that is used in the treatment of RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Tunisia (3):
  - Sfax
  - Sousse
  - Tunis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenous infusion once every 4 weeks, for a total of 6 infusions during the initial phase of the study. Participants who completed the initial phase and had at least one moderate response according to the European League Against Rheumatism (EULAR) category entered the extension phase and received an additional 6 infusions of 8 mg/kg tocilizumab every 4 weeks.
Period: Initial Phase
Arm/Group | Tocilizumab
Started | 51
Completed | 46
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Pregnancy | 1
Period: Extension Phase
Arm/Group | Tocilizumab
Started | 45 (1 participant withdrew consent after completing initial phase and did not enter the extension phase)
Completed | 41
Not Completed | 4
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received at least one dose of medication and for whom at least one post baseline safety measurement was available.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg intravenous infusion once every 4 weeks, for a total of 6 infusions during the initial phase of the study. Participants who completed the initial phase and had at least one moderate response according to the EULAR category entered the extension phase and received an additional 6 infusions of 8 mg/kg tocilizumab every 4 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.01 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 5

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieved Clinically Significant Improvement Assessed Using Disease Activity Score Based on 28 Joints (DAS28)
Description: DAS28 calculated from the swollen joint count (SJC) and tender joint count (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and participant's global assessment (PtGA) of disease activity by Visual analog Scale (VAS; participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 less than or equal to (≤) 3.2 equals (=) low disease activity (LDA), DAS28 greater than (>) 3.2 to 5.1 = moderate to high disease activity. A reduction of at least 1.2 units in DAS28 was considered clinically significant improvement.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; number (n)= number of participants analyzed at a specific visit
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  Week 4 (n=51) | 56.9
  Week 8 (n=49) | 81.6
  Week 12 (n=47) | 83.0
  Week 16 (n=47) | 80.9
  Week 20 (n=46) | 95.7
  Week 24 (n=46) | 91.3
  Week 36 (n=43) | 86.0
  Week 48 (n=41) | 92.7
  Week 52 (n=42) | 90.5

2. Secondary Outcome: Percentage of Participants Achieving LDA Assessed Using DAS28
Description: DAS28 calculated from the SJC and TJC using the 28 joints count, the ESR (mm/hour) and PtGA of disease activity (VAS) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 less than (<) 3.2 = LDA.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants analyzed at a specific visit
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  Week 4 (n=51) | 9.8
  Week 8 (n=49) | 26.5
  Week 12 (n=47) | 34.0
  Week 16 (n=47) | 36.2
  Week 20 (n=46) | 52.2
  Week 24 (n=46) | 47.8
  Week 36 (n=43) | 55.8
  Week 48 (n=41) | 65.9
  Week 52 (n=42) | 61.9

3. Secondary Outcome: Percentage of Participants Achieving Remission Assessed Using DAS28
Description: DAS28 calculated from the SJC and TJC using the 28 joints count, the ESR (mm/hour) and PtGA of disease activity (VAS) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. Participants were considered in remission when reaching a DAS28 score <2.6.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants analyzed at a specific visit
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  Baseline (n=51) | 0.0
  Week 4 (n=51) | 2.0
  Week 8 (n=49) | 12.2
  Week 12 (n=47) | 23.4
  Week 16 (n=47) | 23.4
  Week 20 (n=46) | 32.6
  Week 24 (n=46) | 41.3
  Week 36 (n=43) | 44.2
  Week 48 (n=41) | 41.5
  Week 52 (n=42) | 45.2

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Percent (%), 50% or 70% Improvement (ACR20/ACR50/ACR70)
Description: The ACR response rates ACR20/ACR50/ACR70 are defined as ≥20%, ≥50%, or ≥70% improvement, respectively, in SJC and TJC, as well as a ≥20%, ≥50%, or ≥70% improvement, respectively, in 3 of the 5 remaining core ACR assessments: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a Health Assessment Questionnaire (HAQ), and 5) C-reactive protein (CRP) at each visit.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  Week 4 ACR20 | 29.2
  Week 4 ACR50 | 6.3
  Week 4 ACR70 | 0.0
  Week 8 ACR20 | 54.3
  Week 8 ACR50 | 21.7
  Week 8 ACR70 | 4.3
  Week 12 ACR20 | 61.2
  Week 12 ACR50 | 32.7
  Week 12 ACR70 | 12.2
  Week 16 ACR20 | 49.0
  Week 16 ACR50 | 24.5
  Week 16 ACR70 | 18.4
  Week 20 ACR20 | 70.8
  Week 20 ACR50 | 35.4
  Week 20 ACR70 | 12.5
  Week 24 ACR20 | 66.7
  Week 24 ACR50 | 33.3
  Week 24 ACR70 | 13.7
  Week 36 ACR20 | 54.2
  Week 36 ACR50 | 33.3
  Week 36 ACR70 | 14.6
  Week 48 ACR20 | 66.0
  Week 48 ACR50 | 48.9
  Week 48 ACR70 | 27.7
  Week 52 ACR20 | 58.3
  Week 52 ACR50 | 37.5
  Week 52 ACR70 | 18.8

5. Secondary Outcome: Time To Achieve ACR20/ACR50/ACR70
Description: The ACR response rates ACR20/ACR50/ACR70 are defined as ≥20%, ≥50%, or ≥70% improvement, respectively, in SJC and TJC, as well as a ≥20%, ≥50%, or ≥70% improvement, respectively, in 3 of the 5 remaining core ACR assessments: 1) physician's global assessment of disease activity, 2) participant's assessment of disease activity, 3) participant's assessment of pain, 4) participant's assessment of functional disability via (HAQ, and 5) CRP at each visit. The median time to achieve ACR20/ACR50/ACR70 was calculated using Kaplan-Meier estimates.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
weeks
  ACR20 | 8.0 [4.0 to 20.0]
  ACR50 | 20.0 [12.0 to NA] — Calculation was not possible due to the small number of participants achieving ACR50
  ACR70 | NA [20.0 to NA] — Calculation was not possible due to the small number of participants achieving ACR70

6. Secondary Outcome: SJC and TJC
Description: 28 joints were assessed for swelling and tenderness. Joints were classified as swollen (1)/not swollen (0) and tender (1)/not tender (0) giving a total possible SJC and TJC score of 0 to 28 each.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
joints
  Baseline TJC (n=51) | 14.3 [12.3 to 16.4]
  Baseline SJC (n=51) | 7.0 [5.7 to 8.2]
  Week 4 TJC (n=51) | 10.3 [8.1 to 12.4]
  Week 4 SJC (n=51) | 5.2 [3.9 to 6.5]
  Week 8 TJC (n=46) | 5.0 [3.8 to 6.3]
  Week 8 SJC (n=49) | 3.4 [2.5 to 4.3]
  Week 12 TJC (n=47) | 5.1 [3.6 to 6.6]
  Week 12 SJC (n=47) | 2.6 [1.7 to 3.4]
  Week 16 TJC (n=47) | 4.7 [3.1 to 6.2]
  Week 16 SJC (n=47) | 3.1 [1.9 to 4.4]
  Week 20 TJC (n=46) | 3.4 [2.4 to 4.3]
  Week 20 SJC (n=46) | 1.6 [1.1 to 2.2]
  Week 24 TJC (n=46) | 3.5 [2.2 to 4.9]
  Week 24 SJC (n=46) | 1.6 [0.8 to 2.4]
  Week 28 TJC (n=34) | 3.3 [2.3 to 4.3]
  Week 28 SJC (n=34) | 1.3 [0.7 to 2.0]
  Week 32 TJC (n=34) | 2.5 [1.8 to 3.3]
  Week 32 SJC (n=34) | 1.4 [0.7 to 2.1]
  Week 36 TJC (n=41) | 3.6 [2.1 to 5.0]
  Week 36 SJC (n=41) | 2.0 [1.2 to 2.8]
  Week 40 TJC (n=33) | 2.6 [1.7 to 3.6]
  Week 40 SJC (n=33) | 1.3 [0.5 to 2.0]
  Week 44 TJC (n=34) | 2.6 [1.4 to 3.8]
  Week 44 SJC (n=34) | 1.5 [0.7 to 2.4]
  Week 48 TJC (n=39) | 2.4 [1.4 to 3.4]
  Week 48 SJC (n=39) | 1.2 [0.7 to 1.7]
  Week 52 TJC (n=40) | 2.8 [1.4 to 4.2]
  Week 52 SJC (n=40) | 1.9 [1.2 to 2.7]

7. Secondary Outcome: Assessment of Pain by the Participant Using Visual Analog Scale (VAS)
Description: The participants assessed their pain using a 0 to 100 millimeter (mm) horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". The participants marked the line corresponding to their level of pain and the distance from the left edge was measured.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
mm
  Baseline (n=50) | 67.6 [62.5 to 72.6]
  Week 4 (n=48) | 49.4 [43.8 to 55.0]
  Week 8 (n=47) | 40.6 [35.3 to 46.0]
  Week 12 (n=47) | 36.0 [30.5 to 41.5]
  Week 16 (n=48) | 36.1 [30.8 to 41.4]
  Week 20 (n=45) | 33.2 [27.8 to 38.5]
  Week 24 (n=46) | 28.5 [23.6 to 33.3]
  Week 36 (n=44) | 30.0 [23.1 to 36.9]
  Week 48 (n=41) | 22.9 [15.9 to 29.9]
  Week 52 (n=40) | 23.7 [17.4 to 30.0]

8. Secondary Outcome: Assessment of Global Disease by the Participant Using VAS
Description: The participant's global assessment of disease activity was assessed using a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). The participants marked the line corresponding to their assessment of disease activity and the distance from the left edge was measured.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
mm
  Baseline (n=51) | 64.7 [59.6 to 69.7]
  Week 4 (n=51) | 52.9 [46.0 to 59.9]
  Week 8 (n=48) | 40.9 [36.2 to 45.6]
  Week 12 (n=47) | 37.1 [32.0 to 42.2]
  Week 16 (n=48) | 34.4 [28.7 to 40.0]
  Week 20 (n=45) | 32.6 [27.2 to 38.0]
  Week 24 (n=46) | 29.3 [24.3 to 34.4]
  Week 36 (n=44) | 28.7 [21.8 to 35.6]
  Week 48 (n=41) | 20.1 [14.6 to 25.5]
  Week 52 (n=41) | 24.1 [17.9 to 30.4]

9. Secondary Outcome: Assessment of Global Disease by the Physician Using Visual Analog Scale (VAS)
Description: The physician's global assessment of disease activity was assessed using a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). The physician marked the line corresponding to their assessment of disease activity and the distance from the left edge was measured.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
mm
  Baseline (n=51) | 58.8 [54.0 to 63.6]
  Week 4 (n=51) | 45.9 [41.1 to 50.7]
  Week 8 (n=48) | 35.5 [31.6 to 39.4]
  Week 12 (n=47) | 31.1 [26.7 to 35.5]
  Week 16 (n=48) | 32.3 [26.9 to 37.8]
  Week 20 (n=45) | 28.9 [24.0 to 33.9]
  Week 24 (n=46) | 26.4 [21.6 to 31.3]
  Week 36 (n=44) | 23.5 [17.8 to 29.2]
  Week 48 (n=41) | 19.6 [14.8 to 24.5]
  Week 52 (n=40) | 19.6 [14.8 to 24.4]

10. Secondary Outcome: Assessment of Physical Function Using Health Assessment Questionnaire (HAQ)
Description: Physical function was assessed using the HAQ. The HAQ scores range from 0 to 3 with, 0: no assistance needed, 1: participant uses a special device for day-to-day activities, 2: participant usually needs help from another person, and 3: participant uses BOTH a special device AND another person's help for day-to-day activities.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
units on a scale
  Baseline (n=51) | 1.7 [1.5 to 1.9]
  Week 4 (n=50) | 1.2 [1.0 to 1.4]
  Week 8 (n=48) | 1.7 [0.6 to 2.7]
  Week 12 (n=47) | 0.9 [0.7 to 1.1]
  Week 16 (n=48) | 0.8 [0.6 to 1.0]
  Week 20 (n=46) | 0.8 [0.6 to 1.0]
  Week 24 (n=46) | 0.7 [0.6 to 0.9]
  Week 36 (n=40) | 1.0 [0.6 to 1.4]
  Week 48 (n=37) | 0.9 [0.6 to 1.1]
  Week 52 (n=38) | 0.8 [0.6 to 1.0]

11. Secondary Outcome: Mean C-Reactive Protein (CRP) Levels
Description: CRP is an acute phase reactant and levels of CRP increase with inflammation. CRP is measured as milligrams per liter (mg/L).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
mg/L
  Baseline (n=51) | 26.6 [18.4 to 34.8]
  Week 4 (n=51) | 10.4 [4.9 to 15.9]
  Week 8 (n=49) | 9.5 [4.3 to 14.6]
  Week 12 (n=47) | 8.4 [4.7 to 12.1]
  Week 16 (n=46) | 9.1 [4.7 to 13.5]
  Week 20 (n=46) | 10.9 [5.9 to 15.9]
  Week 24 (n=44) | 11.0 [5.1 to 16.8]
  Week 36 (n=43) | 12.4 [2.1 to 22.7]
  Week 48 (n=42) | 10.4 [4.3 to 16.4]
  Week 52 (n=40) | 7.4 [4.3 to 10.5]

12. Secondary Outcome: Mean Erythrocyte Sedimentation Rate (ESR) Levels
Description: ESR is an acute phase reactant and levels of ESR increase with inflammation. ESR is measured as mm/hour.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 36, 48 and 52
Population: Safety population; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (95% Confidence Interval); unit: mm/hour
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
mm/hour
  Baseline (n=51) | 44.1 [35.7 to 52.4]
  Week 4 (n=51) | 21.0 [13.2 to 28.9]
  Week 8 (n=49) | 22.1 [12.8 to 31.4]
  Week 12 (n=47) | 17.0 [12.4 to 21.7]
  Week 16 (n=47) | 16.8 [11.5 to 22.0]
  Week 20 (n=46) | 13.5 [9.2 to 17.8]
  Week 24 (n=46) | 18.4 [12.3 to 24.5]
  Week 36 (n=43) | 15.6 [9.2 to 22.0]
  Week 48 (n=42) | 17.7 [11.8 to 23.6]
  Week 52 (n=42) | 16.9 [11.2 to 22.6]

13. Secondary Outcome: Percentage of Participants Experiencing Fatigue
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: Safety population; n=number of participants analyzed for the given parameter at the specified visit
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  Baseline (n=50) | 22.0
  Week 4 (n=49) | 16.3
  Week 8 (n=48) | 4.2
  Week 12 (n=45) | 13.3
  Week 16 (n=47) | 10.6
  Week 20 (n=44) | 11.4
  Week 24 (n=46) | 10.9

14. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious AEs (SAEs), Related AEs, Discontinuation Due to AEs, or Death
Time Frame: Baseline, every 4 weeks through Week 52
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
percentage of participants
  AEs | 78.4
  SAEs | 5.9
  Related AEs | 15.2
  Discontinuation due to AE | 7.8
  Death | 0

15. Secondary Outcome: Number of Participants Who Discontinued Tocilizumab
Time Frame: Week 52
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 51
participants | 1

ADVERSE EVENTS:
Time Frame: AEs were recorded from the date of first infusion until the end of study at 52 weeks.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 3/51
Other Adverse Events (participants affected / at risk) | 39/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=51)
Confusional syndrome (Nervous system disorders) | 1
Whitlows of the toe (Surgical and medical procedures) | 1
Pleural-pneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=51)
Oral ulcer (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Acute appendicitis (Surgical and medical procedures) | 1
Osteoarticular fracture (fifth metatarsal) (Musculoskeletal and connective tissue disorders) | 1
Osteomalacia (Musculoskeletal and connective tissue disorders) | 1
Skin and subcutaneous lesions (Skin and subcutaneous tissue disorders) | 8
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Flu syndrome (General disorders) | 3
Urinary infection (Renal and urinary disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Increased ALT/AST (Investigations) | 15
Hypercholesterolemia (Investigations) | 18
Hypertriglyceridemia (Investigations) | 17
Neutropenia (Investigations) | 8
Cytolysis (Investigations) | 1
Reticulocytosis (Investigations) | 1
Oral thrush (Infections and infestations) | 1
Headache (General disorders) | 1
Dizziness (Ear and labyrinth disorders) | 2
Asthenia (General disorders) | 1
Erythematous plaque of Elbows (Skin and subcutaneous tissue disorders) | 1
Hiatal hernia esopahgitis (Gastrointestinal disorders) | 1
Erythematous purpuric lesions (Skin and subcutaneous tissue disorders) | 1
Papular skin lesions (Skin and subcutaneous tissue disorders) | 3
Hyperbilirubinemai (Hepatobiliary disorders) | 2
Lower gastrointestinal bleeding - Hemorrhoids (Gastrointestinal disorders) | 1
Vasodilation of feet (General disorders) | 1
Hyperisonophilia (Blood and lymphatic system disorders) | 1
Hypokalemia (General disorders) | 1
Hallux Abscess (General disorders) | 1
Bronchial Infectious syndrome (Infections and infestations) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Epigastric pain (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.